CLINICAL TRIAL: NCT04301414
Title: A Pilot Study of Neoadjuvant Non-fucosylated Anti-CTLA-4 (BMS-986218) + Degarelix Acetate vs. Degarelix Acetate Alone in Men With High-risk Localized Prostate Cancer
Brief Title: Non-fucosylated Anti-CTLA-4 (BMS-986218) + Degarelix Acetate vs. Degarelix Acetate Alone in Men With High-risk Localized Prostate Cancer
Acronym: Neo-Red-P
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Karie D. Runcie, MD, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAS3560
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety lead-in (Other): The first 4 subjects enrolled will be given degarelix plus BMS-986218.
  Interventions: Drug: BMS-986218 and Degarelix
- Arm A (Active Comparator): Degarelix 240mg subcutaneous (SQ) x1 dose 2 weeks prior to radical prostatectomy
  Interventions: Drug: Degarelix
- Arm B (Experimental): BMS-986218 20mg IV every 2 weeks x 2 doses starting 3 weeks prior to radical prostatectomy plus degarelix 240mg SQ x1 dose 2 weeks prior to radical prostatectomy.
  Interventions: Drug: BMS-986218 and Degarelix

INTERVENTIONS:
Drug: BMS-986218 and Degarelix — BMS-986218 20mg IV every 2 weeks x 2 doses starting 3 weeks prior to radical prostatectomy plus degarelix 240mg subcutaneous (SQ) x1 dose 2 weeks prior to radical prostatectomy.
  Arms: Arm B; Safety lead-in
Drug: Degarelix — Degarelix 240mg SQ x1 dose 2 weeks prior to radical prostatectomy
  Arms: Arm A

SUMMARY:
The purpose of this study is to see whether immunotherapy with BMS-986218 added to degarelix (which suppresses testosterone) given prior to surgery can decrease the chance that cancer will come back compared to degarelix alone. People who usually have this type of prostate cancer usually do not receive any additional therapy prior to surgery. Approximately 24 individuals will be asked to participate in this study.

DETAILED DESCRIPTION:
This is a single-center, randomized, two-arm, study evaluating the safety, feasibility and immunogenicity of neoadjuvant degarelix(Arm A) or BMS-986218 plus degarelix (Arm B) prior to radical prostatectomy in men with high-risk localized prostate cancer (neo-RED-P). Our primary objective is to characterize safety, tolerability, and feasibility of degarelix with or without BMS-986218 in the neoadjuvant setting. The trial will monitor toxicity and safety, as well as surgery related adverse events. The secondary objectives will be to evaluate an immune response consistent with the proposed mechanism of action of BMS-986218, depletion of Tregs, and to assess the pathologic complete response rate, PSA response rate and time-to-PSA recurrence following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (clinical stage T1c-T3b, N0, M0) without involvement of lymph nodes, bone, or visceral organs
* Initial prostate biopsy is available for central pathologic review, and is confirmed to show at least 2 positive cores and a Gleason sum of ≥4+3
* Radical prostatectomy has been scheduled at Columbia University Irving Medical Center
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1, or Karnofsky score ≥ 70% (see Appendix A)
* Adequate bone marrow, hepatic, and renal function:

  * White blood cell count (WBC) >3,000 cells/mm3
  * Absolute neutrophil count (ANC)>1,500 cells/mm3
  * Hemoglobin >9.0 g/dL
  * Platelet count >100,000 cells/mm3
  * Serum creatinine <1.5 × upper limit of normal (ULN)
  * Serum bilirubin <1.5 × ULN
  * Alanine transaminase (ALT) <3 × ULN
  * Aspartate aminotransferase (AST)<3 × ULN
  * Alkaline phosphatase <3 × ULN
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent)
* Willingness to use barrier contraception from the time of first dose of BMS-986218 until 165 days from the last dose of BMS-986218.

Exclusion Criteria:

* Presence of known lymph node involvement or distant metastases
* Other histologic types of prostate cancers such as ductal, sarcomatous, lymphoma, small cell, and neuroendocrine tumors
* Prior radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for prostate cancer
* Prior immunotherapy/vaccine therapy for prostate cancer
* Concomitant treatment with other hormonal therapy or 5α-reductase inhibitors (prior use of these agents is allowed).
* Conditions requiring systemic treatment with either corticosteroids > 10 mg daily prednisone equivalents or other immunosuppressive medications within 14 days of study treatment administration, except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease.

  (1) Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted.
* History of known or suspected autoimmune disease with the following exceptions:

  * Vitiligo
  * Resolved childhood atopic dermatitis
  * Psoriasis (with exception of psoriatic arthritis) not requiring systemic treatment (within the past 2 years).
  * Patients with Grave's disease or Hashimoto's thyroiditis that are now euthyroid clinically and by laboratory testing.
* History of malignancy within the last 2 years, with the exception of non-melanoma skin cancers and superficial bladder cancer
* Known uncontrolled or significant cardiovascular disease including, but not limited, to any of the following:

  1. Myocardial infarction or stroke/transient ischemic attack within the past 6 months.
  2. Uncontrolled angina within the past 3 months.
  3. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes).
  4. History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, or significant pericardial effusion).
  5. History of myocarditis, regardless of etiology.
  6. Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
* Known prior or current history of HIV.
* Patients with known untreated hepatitis B/C or those with a detectable viral load.
* Active infection ≤7 days prior to start of treatment.
* Live vaccine within 30 days of start of treatment.
* Prior history of hypersensitivity to a monoclonal antibody.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with an adverse event will be reported with an exact binomial 95% confidence interval | 42 months
  Characterizing the safety, tolerability, and feasibility of degarelix with or without BMS-986218 in the neoadjuvant setting. All subjects receiving at least one dose of the study drug(s) will be evaluable for toxicity.

SECONDARY OUTCOMES:
Mean Treg cell staining percentage in harvested prostate tissues will be reported and compared post-treatment between the treatment groups using paired sample test. | 42 months
  The standard deviation, 95% confidence interval, median, and range of values will also be reported where appropriate
Pathological complete responses (pCR)- an absence of tumor identification on standard histological analysis of the resected prostate specimens. | 42 months
  The estimate and 95% confidence intervals will be obtained.
Undetectable PSA at 12 months- the proportion of patients who achieve an undetectable PSA (<0.1 ng/mL) by 12 months after prostatectomy | 42 months
  The estimate and 95% confidence intervals will be obtained.
PSA response rates- a 50% change in pre-treatment and post-treatment PSA. | 42 months
  These endpoints will be expressed as the proportion of men achieving a PSA response. The estimate and 95% confidence intervals will be obtained.
Time to PSA recurrence- the interval from the time of prostatectomy to the time when the first of at least two serial rises in PSA (≥2 weeks apart) with a PSA ≥0.2 ng/mL. | 42 months
  PSA will be measured every 3 (±1) months during the first post-operative year and every 6 (±2) months during the second and third post-operative years. For subjects who have not yet demonstrated PSA relapse after 3 years followup patients will be censored at the date of the last assessment that shows a lack of PSA recurrence. This outcome will be expressed as a median (95% CI) and will be determined using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Karie D. Runcie, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided